CLINICAL TRIAL: NCT05367063
Title: Canagliflozin Attenuates CMR-Quantified Myocardial Fibrosis in Patients With Type 2 Diabetes Mellitus at High Cardiovascular Risk
Brief Title: Canagliflozin and Myocardial Fibrosis
Acronym: CANA-DIA-FIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSE-202112
Record Dates: First submitted 2021-12-07; First posted 2022-05-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Cardiovascular Risk
Keywords: SGLT2 inhibitor; Canagliflozin; Type 2 diabetes mellitus; Myocardial fibrosis; Cardiac magnetic resonance; Cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: On the basis of a stable dose of metformin, the test group was treated with Canagliflozin tablets (SGLT2 inhibitor), and the control group was treated with Sitagliptin tablets (DPP-4 inhibitor).
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluators only know the subjects' numbers and have no knowledge of other clinical information about the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canagliflozin group (Active Comparator): On the basis of the original metformin medication, the experimental group took canagliflozin 1 tablet (100 mg) orally once a day (qd) before the first meal of the day, and the dosing cycle lasts 6 months.
  Interventions: Drug: Canagliflozin 100mg or Sitagliptin 100mg
- Sitagliptin group (Placebo Comparator): On the basis of the original metformin medication, the experimental group took Sitagliptin 1 tablet (100 mg) orally once a day (qd) before the first meal of the day, and the dosing cycle lasts 6 months.
  Interventions: Drug: Canagliflozin 100mg or Sitagliptin 100mg

INTERVENTIONS:
Drug: Canagliflozin 100mg or Sitagliptin 100mg — Eligible type 2 diabetes patients at high risks of cardiovascular diseases will be randomly assigned by a 1:1 ratio to either Canagliflozin 100 mg once daily or Sitagliptin 100 mg once daily.

SUMMARY:
Recently, large clinical intervention studies have demonstrated the cardiovascular protective effects on of sodium-glucose cotransporter 2 inhibitors (SGLT2i) such as empagliflozin, dapagliflozin, and canagliflozin in reduction of cardiovascular and all-cause mortality, coincident with a significant reduction in heart failure hospitalizations. Therefore, SGLT2i had been recommended as a therapeutic drug for diabetic patients to reduce the occurrence of cardiovascular events. However, the mechanism of these benefits remains unclear at the present time.

Myocardial fibrosis is not only an important physiopathological mechanism of heart failure, but also has been shown to be closely associated with the risk of heart failure-related hospitalization and death, especially in patients with T2D. However, whether SGLT2i can exert cardioprotective effects by improving myocardial fibrosis remains to be further investigated. In recent years, the development of cardiac magnetic resonance (CMR) technology enables to detect focal and diffuse fibrosis in myocardial tissue, which makes it possible to systematically explore the role of SGLT2i on myocardial fibrosis. Although several studies including EMPA-HEART, SUGAR-DM-HF have explored the effects of SGLT2i on cardiac structure and function, these studies didn't reach consistent results. In addition, more scarce studies have investigated the effects of SGLT2i on both focal and diffuse fibrosis. At present, whether SGLT2i treatment can change the relevant indicators of myocardial fibrosis in people with diabetes and cardiovascular risk factors has not yet been reported. In addition, previous studies mainly focus on empagliflozin and dapagliflozin, and studies on canagliflozin are still very scarce. Therefore, this study intends to explore the effects of canagliflozin on myocardial fibrosis and other structures and functions of the heart in patients with type 2 diabetes mellitus and high cardiovascular risk factors.

DETAILED DESCRIPTION:
According to the International Federation for Diabetes, diabetes now affects approximately 9.3% of the population worldwide, and the prevalence over the next two decades will continue to increase, reaching 552 million by 2030. In particular, type 2 diabetes (T2D) can cause macrovascular and microvascular complications, for example, T2D can increase the risks of ischemic stroke by 72% and stable angina by 62%. In addition, the incidence of heart failure in T2D patients is 9-22%, 2-4 times that of the general population. A significant breakthrough in contemporary cardiology was the finding that sodium-glucose-cotransporter-2 (SGLT2) inhibitors are associated with a lower risk of heart failure (HF) Hospitalization in patients with or at high risk of CV disease. In the EMPAREG OUTCOME Trial, Empagliflozin reduced cardiovascular death and hospitalisation for heart failure (HF) by 38% and 35%, respectively, with an almost immediate beneficial effect despite only a modest difference in glycaemic control, comparing two study arms over 94 weeks. The reductions in CV death were not accounted for by the reductions in atherothrombotic outcomes, as the rates of myocardial infarction and stroke remained unchanged with therapy. The proposed theory that HF is the outcome most sensitive to SGLT2 inhibition was confirmed in the Canagliflozin Cardiovascular Assessment Study (CANVAS) Program and Dapagliflozin DECLARE-TIMI 58 trials. More recently, the EMPEROR trial showed that SGLT2 inhibition reduces the risk of hospitalisation for HF in patients regardless of the presence or absence of diabetes. The mechanisms by which SGLT2 inhibitors cause the reduction in HF risks and cardiovascular mortality are yet unknown.

Myocardial fibrosis is not only an important physiopathological mechanism of heart failure, but also has been shown to be closely associated with the risk of heart failure-related hospitalization and death, especially in patients with T2D. However, whether SGLT2i can exert cardioprotective effects by improving myocardial fibrosis remains to be further investigated. In recent years, the development of cardiac magnetic resonance (CMR) technology enables to detect focal and diffuse fibrosis in myocardial tissue, which makes it possible to systematically explore the role of SGLT2i on myocardial fibrosis.

At present, relevant studies have explored the effects of SGLT2i on cardiac structure and function. For example, there have been several related studies on left ventricular structure and function, but no consistent conclusions have been drawn: for example, the EMPA-HEART study showed that empagliflozin can reduce left ventricular mass; DAPA-HEART The LVH and SUGAR-DM-HF studies clarified the effect of dapagliflozin in reducing left ventricular mass and end-systolic volume; the REFORM study did not find that dapagliflozin had any effect on left ventricular weight. plastic effect. In addition, only the EMPA-HEART study investigated the effect of SGLT2i on both focal and diffuse fibrosis, and found that empagliflozin significantly improved diffuse fibrosis in people with diabetes and coronary heart disease. However, the SUGAR-DM-HF study did not observe changes in diffuse fibrosis with empagliflozin intervention in people with diabetes or prediabetes with reduced ejection fraction. At present, whether SGLT2i treatment can change the relevant indicators of myocardial fibrosis in people with diabetes and cardiovascular risk factors has not yet been reported. In addition, previous studies mainly focus on empagliflozin and dapagliflozin, and studies on canagliflozin are still very scarce. Therefore, this study intends to explore the effects of canagliflozin on myocardial fibrosis and other structures and functions of the heart in patients with type 2 diabetes mellitus and high cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes;
* Haemoglobin A1c ≥7.0% and < 10.5%;
* Patients who have received a stable dose of metformin or metformin combined with insulin secretagogues and/or insulin therapy for 4 weeks before enrollment;
* Those who met at leat one of the following criteria:

  1. Patients with at least 3 of the folllowing risk factors: (1) male >55 years old, or female > 65 years old; (2) BMI≥25 kg/m2; (3) hypertension; (4) dyslipidemia; (5) current smoker (Brinkman index ≥ 200;
  2. Any of the following signs of target organ damage are present: (1) albuminuria (ACR≥300mg/g); (2) 45 ml/min/1.73 m2 ≤eGFR<90 ml/ min/1.73 m2; (3) Left ventricular hypertrophy or coupled with retinopathy.

Exclusion Criteria:

* Female subjects who are pregnant, lactating or of child bearing potential, or pre-menopausal women. (Menopause will be determined by patient and physician history;
* Subjects currently treated with SGLT2 inhibitors, GLP1 receptor agonist, or sitagliptin;
* Significant allergy or known intolerance to Canagliflozin or Sitagliptin;
* History of hypovolemia, amputation, peripheral vascular disease, diabetic foot ulcers;
* History of diagnosed cardiovascular diseases, including myocardial infarction, hospitalization for unstable angina pectoris, cerebral infarction (ischemic stroke), coronary artery bypass grafting, percutaneous coronary intervention (with or without stents) Implantation), peripheral vascular reconstruction (angioplasty or surgery), heart failure, arrhythmia, heart valve disease;
* AST or ALT ≥ 3 times the upper limit of normal;
* eGFR <45 ml/min/1.73 m2；
* type 1 diabetes;
* Diabetic ketosis or diabetic hyperosmolar coma;
* History of respiratory disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension, etc.);
* Existing hypertensive emergency (systolic/diastolic blood pressure exceeding 180/120mmHg) at the time of enrollment, or evaluated For refractory hypertension (after the use of sufficient doses of 3 antihypertensive drugs, the systolic blood pressure is still> 140 or Diastolic blood pressure> 90mmHg);
* Known impaired gastrointestinal function or gastrointestinal diseases that may significantly affect the absorption of the test drug, such as: diagnosed active ulcers (Forrest grade II and below), inflammatory bowel disease, malabsorption related diseases, and non-absorbent diseases. Controlled diarrhea, gastrointestinal surgery (such as bariatric surgery);
* Patients with diagnosed malignant tumors;
* Participate in other clinical trials within 3 months;
* Other creteria that were not eligible to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in myocardial fibrosis | 26 weeks since the randomization
  The rate of ventricular extracellular volume and late gadolinium enhancement measured by MRI

SECONDARY OUTCOMES:
Change in Left Ventricle (LV) Structure/Function | 26 weeks since the randomization
  1. Change in left ventricle end-diastolic volume (LVEDV) and index (LVEDVI), left ventricle end-systolic volume (LVESV) and index (LVESVI), and left ventricle ejection fraction (LVEF) , measured by CMR.
  2. Change in left ventricular end-diastolic/systolic diameter (LVEDD/LVESD), left ventricular ejection fraction (LVEF), interventricular septal thickness (IVS), left ventricular posterior wall thickness (LVPW), left atrial anteroposterior diameter (LA), aortic root dimension at the sinus of Valsalva (AORD), and pulmonary artery systolic pressure (PASP), measured by Echocardiography.
Change in resting mocardial blood flow | 26 weeks since the randomization
  The rate of resting myocardial blood flow (MBF, ml/min) measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: SAP
Time Frame: No time limited.
Access Criteria: Anyone can access the Statistical Analysis Plan (SAP).
URL: https://register.clinicaltrials.gov/e307c484-addf-4c15-be07-9a2e4dc11afc

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Emerging Risk Factors Collaboration; Di Angelantonio E, Kaptoge S, Wormser D, Willeit P, Butterworth AS, Bansal N, O'Keeffe LM, Gao P, Wood AM, Burgess S, Freitag DF, Pennells L, Peters SA, Hart CL, Haheim LL, Gillum RF, Nordestgaard BG, Psaty BM, Yeap BB, Knuiman MW, Nietert PJ, Kauhanen J, Salonen JT, Kuller LH, Simons LA, van der Schouw YT, Barrett-Connor E, Selmer R, Crespo CJ, Rodriguez B, Verschuren WM, Salomaa V, Svardsudd K, van der Harst P, Bjorkelund C, Wilhelmsen L, Wallace RB, Brenner H, Amouyel P, Barr EL, Iso H, Onat A, Trevisan M, D'Agostino RB Sr, Cooper C, Kavousi M, Welin L, Roussel R, Hu FB, Sato S, Davidson KW, Howard BV, Leening MJ, Leening M, Rosengren A, Dorr M, Deeg DJ, Kiechl S, Stehouwer CD, Nissinen A, Giampaoli S, Donfrancesco C, Kromhout D, Price JF, Peters A, Meade TW, Casiglia E, Lawlor DA, Gallacher J, Nagel D, Franco OH, Assmann G, Dagenais GR, Jukema JW, Sundstrom J, Woodward M, Brunner EJ, Khaw KT, Wareham NJ, Whitsel EA, Njolstad I, Hedblad B, Wassertheil-Smoller S, Engstrom G, Rosamond WD, Selvin E, Sattar N, Thompson SG, Danesh J. Association of Cardiometabolic Multimorbidity With Mortality. JAMA. 2015 Jul 7;314(1):52-60. doi: 10.1001/jama.2015.7008. PMID 26151266
- [Background] Dunlay SM, Givertz MM, Aguilar D, Allen LA, Chan M, Desai AS, Deswal A, Dickson VV, Kosiborod MN, Lekavich CL, McCoy RG, Mentz RJ, Pina IL; American Heart Association Heart Failure and Transplantation Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and the Heart Failure Society of America. Type 2 Diabetes Mellitus and Heart Failure: A Scientific Statement From the American Heart Association and the Heart Failure Society of America: This statement does not represent an update of the 2017 ACC/AHA/HFSA heart failure guideline update. Circulation. 2019 Aug 13;140(7):e294-e324. doi: 10.1161/CIR.0000000000000691. Epub 2019 Jun 6. PMID 31167558
- [Background] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Background] Hudsmith LE, Petersen SE, Tyler DJ, Francis JM, Cheng AS, Clarke K, Selvanayagam JB, Robson MD, Neubauer S. Determination of cardiac volumes and mass with FLASH and SSFP cine sequences at 1.5 vs. 3 Tesla: a validation study. J Magn Reson Imaging. 2006 Aug;24(2):312-8. doi: 10.1002/jmri.20638. PMID 16795076
- [Background] Verma S, Mazer CD, Yan AT, Mason T, Garg V, Teoh H, Zuo F, Quan A, Farkouh ME, Fitchett DH, Goodman SG, Goldenberg RM, Al-Omran M, Gilbert RE, Bhatt DL, Leiter LA, Juni P, Zinman B, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The EMPA-HEART CardioLink-6 Randomized Clinical Trial. Circulation. 2019 Nov 19;140(21):1693-1702. doi: 10.1161/CIRCULATIONAHA.119.042375. Epub 2019 Aug 22. PMID 31434508
- [Background] Brown AJM, Gandy S, McCrimmon R, Houston JG, Struthers AD, Lang CC. A randomized controlled trial of dapagliflozin on left ventricular hypertrophy in people with type two diabetes: the DAPA-LVH trial. Eur Heart J. 2020 Sep 21;41(36):3421-3432. doi: 10.1093/eurheartj/ehaa419. PMID 32578850
- [Background] Lee MMY, Brooksbank KJM, Wetherall K, Mangion K, Roditi G, Campbell RT, Berry C, Chong V, Coyle L, Docherty KF, Dreisbach JG, Labinjoh C, Lang NN, Lennie V, McConnachie A, Murphy CL, Petrie CJ, Petrie JR, Speirits IA, Sourbron S, Welsh P, Woodward R, Radjenovic A, Mark PB, McMurray JJV, Jhund PS, Petrie MC, Sattar N. Effect of Empagliflozin on Left Ventricular Volumes in Patients With Type 2 Diabetes, or Prediabetes, and Heart Failure With Reduced Ejection Fraction (SUGAR-DM-HF). Circulation. 2021 Feb 9;143(6):516-525. doi: 10.1161/CIRCULATIONAHA.120.052186. Epub 2020 Nov 13. PMID 33186500
- [Background] Singh JSS, Mordi IR, Vickneson K, Fathi A, Donnan PT, Mohan M, Choy AMJ, Gandy S, George J, Khan F, Pearson ER, Houston JG, Struthers AD, Lang CC. Dapagliflozin Versus Placebo on Left Ventricular Remodeling in Patients With Diabetes and Heart Failure: The REFORM Trial. Diabetes Care. 2020 Jun;43(6):1356-1359. doi: 10.2337/dc19-2187. Epub 2020 Apr 3. PMID 32245746

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT05367063/SAP_001.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT05367063/ICF_000.pdf